CLINICAL TRIAL: NCT06611397
Title: Double-Blinded Pilot Feasibility Study of the Discogen Device to Alleviate Discogenic Back/Radicular Leg Pain
Brief Title: Discogen for Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Discogen (Unknown)
Responsible Party: Principal Investigator, Clark Smith, Associate Professor of Rehabilitation and Regenerative Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAU8219
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Disc Herniation
Keywords: Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Treatment Group (Experimental): Study subjects in the treatment group (Arm 1) will receive 3 daily Discogen treatments unilaterally within a one week (M-M) period, each lasting 25 minutes.
  Interventions: Device: Discogen Low pulsed ultrasound treatment
- Sham Control Group (Sham Comparator): Subjects in the sham control arm (Arm 2) will receive 3 daily non-powered treatments unilaterally within a one week (M-M) period, each lasting 25 minutes
  Interventions: Device: Discogen Sham Treatment

INTERVENTIONS:
Device: Discogen Low pulsed ultrasound treatment — The device is a customized Low Intensity Pulsed Ultrasound (LIPUS) transducer system and power source. The transducer is biocompatible for skin contact. The system is capable of calibration to desired treatment parameters. The study subject will be placed in the prone position with all appropriate pressure points padded on the exam table. For the first treatment, fluoroscopic imaging (and/or ultrasonic guidance) will be used to guide the placement of the transducer over the anatomic target, unilateral at the L3-4, L4-5 or L5-S1 levels.
  The skin of the study subject's back will be marked with non-washable marking pen to indicate the site for placing the transducer during the first treatment. The subsequent treatment (second and third) can be done without using ultrasound guidance. The transducer will be placed on the marked site during the second and third treatment.
  The ultrasound signal will be delivered unilaterally for 25 minutes, using a timer visible to the patient. The power ge
  Arms: Treatment Group
Device: Discogen Sham Treatment — The ultrasound signal will be delivered unilaterally for 25 minutes, using a timer visible to the patient. The power generator will not be turned on for the sham treatment, but the wave generator will be displayed. All study subjects will receive a total of three daily Discogen treatments over the span of a single M-M work week
  Arms: Sham Control Group

SUMMARY:
This study will be a double-blinded, two-arm, prospective, randomized controlled pilot feasibility study in 40 evaluable subjects (20 in each arm) at one study site within the United States. Subjects in Arm 1 will receive unilateral Discogen treatment; subjects in Arm 2 will receive unilateral sham treatment (control). Treatment in both arms can include medications, e.g. NSAIDs or muscle relaxants for axial or radicular pain.

DETAILED DESCRIPTION:
This study will be a double-blinded, two-arm, prospective, randomized controlled pilot feasibility study in 40 evaluable subjects (20 in each arm) at one study site within the United States. Subjects in Arm 1 will receive unilateral Discogen treatment; subjects in Arm 2 will receive unilateral sham treatment (control). Treatment in both arms can include medications, e.g. NSAIDs or muscle relaxants for axial or radicular pain. This study will enroll 40 evaluable subjects and follow them for 60 days.

1. Investigate the safety and feasibility of the Discogen device to alleviate back/radicular leg pain
2. Assess the mean reduction in back and radicular leg pain following Discogen treatment.

   * Primary Safety - collection of all adverse events, including any device- or procedure-related adverse events
   * Primary Effectiveness -percent change from baseline for Numerical Pain Scale (NPS) radicular leg pain at 30 and 60 days. The scale ranges from 0(No pain) to 10 (Severe pain).
   * Secondary Effectiveness:

     * Change from baseline in Oswestry Disability Index at 30 and 60 days. The Index ranges from 0-20% (minimal disability), 21-40% (moderate disability), 41-60% (severe disability), 61-80% (crippled), to 81-100% (bed bound).
     * Percent change from baseline NPS back pain at 30 and 60 days

ELIGIBILITY:
Inclusion Criteria

The subject may be included in the study if the following conditions are met:

1. Adult (> 21 y.o.) males and females legally able and willing to participate and provide consent in the study and attend follow-up visits
2. Able and willing to complete study forms and communicate with the investigator
3. Presenting with unilateral radicular leg pain with or without axial back pain of >1 month duration
4. No epidural injections at treatment site within the last three months
5. Leg NPS pain score of 4 - 9 in the last month (on a scale of 0 to 10)
6. Clinical presentation of sensory radiculopathy referable to single-level disc disease/herniation at L3-4, L4-5 or L5-S1
7. MRI lumbar spine negative for extruded disc herniation, tumor, or bleeding, but positive for disc disease/herniation at L3-4, L4-5 or L5-S1 with mild to moderate foraminal or spinal stenosis (less than 50%).

Exclusion Criteria:

1. Pregnant or breastfeeding patient
2. Younger than 21 or older than 75 years
3. Presenting with motor deficits
4. Presenting with a baseline Oswestry Disability Index ≥ 41% (severe disability or worse)
5. Presence of metal hardware within the lumbosacral spine
6. History of spine surgery at the level of treatment.
7. Lumbar spine pathology that may increase procedural risk and/or influence symptoms and/or generate unrelated adverse events (per the discretion of the study PI)
8. Severe lumbar central canal stenosis (greater than 50%)
9. Severe lumbar foraminal stenosis (greater than 50%)
10. Severe herniated lumbar disc 4(Grade 2 and above)
11. Lumbar instability on flexion/extension plain films, greater the Grade 1 spondylolisthesis
12. Unable to understand and complete research questionnaires
13. Any severe medical condition preventing the patient from safely and effectively being treated in the study or reporting study outcomes.
14. BMI greater than 30
15. Implanted spinal stimulators
16. Epidural injections at treatment site within the last three months

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness | 30 and 60 days.
  Percent change from baseline for Numerical Pain Scale (NPS) radicular leg pain at 30 and 60 days. The NPS is a patient-reported assessment of pain intensity, ranging from 0 (No pain) to 10 (Severe pain).
Primary Safety | 60 days
  Collection of all adverse events, including any device or procedure-related adverse events.

SECONDARY OUTCOMES:
Change from baseline in Oswestry Disability Index | 30 and 60 days.
  The Oswestry Disability Index is a patient-reported assessment of level of function (disability) in those living with low back pain. The Index ranges from 0-20% (minimal disability), 21-40% (moderate disability), 41-60% (severe disability), 61-80% (crippled), to 81-100% (bed bound).
Numerical Pain Scale (NPS) | 30 and 60 days.
  Percent change from baseline NPS back pain. The scale ranges from 0 (No pain) to 10 (Severe pain).

CONTACTS AND LOCATIONS:
Overall Officials: Clark Smith, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Su ZH, Liu J, Yang MS, Chen ZY, You K, Shen J, Huang CJ, Zhao QH, Liu EQ, Zhao L, Feng QJ, Pang SM, Li SL, Lu H. Automatic Grading of Disc Herniation, Central Canal Stenosis and Nerve Roots Compression in Lumbar Magnetic Resonance Image Diagnosis. Front Endocrinol (Lausanne). 2022 Jun 6;13:890371. doi: 10.3389/fendo.2022.890371. eCollection 2022. PMID 35733770
- [Background] PASS 2021 Power Analysis and Sample Size Software (2021). NCSS, LLC. Kaysville, Utah, USA, ncss.com/software/pass.
- [Background] Fiore P, Panza F, Cassatella G, Russo A, Frisardi V, Solfrizzi V, Ranieri M, Di Teo L, Santamato A. Short-term effects of high-intensity laser therapy versus ultrasound therapy in the treatment of low back pain: a randomized controlled trial. Eur J Phys Rehabil Med. 2011 Sep;47(3):367-73. Epub 2011 Jun 8. PMID 21654616